CLINICAL TRIAL: NCT05495529
Title: Biliary or Digestive Protection by Room Air Interposition for Thermal Ablation of Central Hepatic Tumors With High Iatrogenic Risk
Brief Title: Biliary or Digestive Protection by Room Air Interposition for Thermal Ablation of Central Hepatic Tumors
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 22Imagerie01
Record Dates: First submitted 2022-08-04; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Radiology, Interventional; Liver Neoplasm; Carcinoma, Hepatocellular (RENI); Neoplasm Metastasis; Ablation Techniques; Radiofrequency Ablation; Microwaves
MeSH Terms: conditions — Liver Neoplasms; Carcinoma; Neoplasm Metastasis | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients with single liver tumor traited by thermoablation with high iatrogenic risk, with biliary or digestive protection by ambiant air interposition
  Interventions: Procedure: Thermal Ablation

INTERVENTIONS:
Procedure: Thermal Ablation — Data collection about complications, succes of the procedure, succes of complete treatement, recurrence, biologic pertubations.

SUMMARY:
This study aims to analyse retrospectively the feasibility, the safety, and the efficiency, of biliary or digestive protection with room air interposition for thermal ablation of central liver tumors with high iatrogenic risk.

Thermal ablation is a mini-invasive and curative treatement of liver tumors. However, it requires to be carefull about surrunding organs, such as digestive structures or central biliary tree, which can be injured if not insulated.

The technique of gas interposition to protect adjacent gut is already known and validated with carbonic gas. Nevertheless, resorption of this gas is very fast, making its use tricky to keep a correct insulation during the whole thermal ablation process.

Room air interposition is easy to use and can offer a slow resorption speed. Furthermore no datas are available concerning the use of room air whatever the organ protected, and the protection of central biliary tree whatever the gas used.

ELIGIBILITY:
Inclusion Criteria :

* Patients with single malignant primary or secondary liver tumor
* Thermal ablation area located within 1 centimeter from central biliary tree or gut
* Thermal insulation using room air interposition
* Follow-up of at least 2 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with single malignant liver tumor with high iatrogenic risk treated by thermal ablation with biliary or digestive protection by room air interposition, in Nice CHU, between January 2013 and December 2021.
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
Feasability | 1 day
  Technical succes of the procedure = feasibility of insulation with room air
Security | 2 months
  Complications (intraoperative clinical or radiological event/abnormality, biological perturbation, clinical event in hospitalization report, imaging request), classified according to SIR (Society of Interventional Radiology) classification in two classes: minor (no additional therapy needed) and major (specific therapy needed) complications.
Efficacity | 2 months
  Response in imaging (MRI or CT) for the tumor treated with thermal ablation
Clinical success | 2 months
  Overall survival

SECONDARY OUTCOMES:
Local and distant recurrence | 2 months
  1. Local recurrence: defined by MRI or CT recurrence within 10 mm from thermal ablation area
  2. Distant recurrence:
  I. Hepatic: defined by MRI or CT intra-hepatic recurrence which is not defined as local recurrence II. Extrahepatic: defined by MRI or CT extra-hepatic recurrence
Local tumorous recurrence free survival | 2 months
  Local tumorous recurrence free survival analysis
Progression free survival | 2 months
  Local or distant recurrence free survival analysis

CONTACTS AND LOCATIONS:
Overall Officials: GARGIULO Manuel, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No